CLINICAL TRIAL: NCT02362464
Title: A Pilot Study of Long Term TARP Vaccination Using A Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccine in Previously Vaccinated Men on NCI 09-C-0139.
Brief Title: Long-Term TARP Vaccination Using a Multi-Epitope TARP Peptide Autologous Dendritic Cell Vaccination in Previously Vaccinated Men on NCI 09-C-0139
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoyoung M. Maeng, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150076; 15-C-0076
Record Dates: First submitted 2015-02-12; First posted 2015-02-13 (Estimated); Results first posted 2022-09-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Neoplasms; Neoplasms of Prostate; Prostate Cancer; Cancer Of Prostate; Stage D0 Prostate Cancer
Keywords: Multi-epitope; Tarp Peptide; Dendritic Cell Vaccine; D0 Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — TARP; Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations (Experimental): Intradermally given vaccine given at weeks 3, 6, 9, 12, 15 and 24.
  Interventions: Biological: Multi-epitope (ME) T-cell Receptor Alternate Reading Frame Protein (TARP) vaccine

INTERVENTIONS:
Biological: Multi-epitope (ME) T-cell Receptor Alternate Reading Frame Protein (TARP) vaccine — dose of 20 x 10^6 viable cells multiepitope TARP dendritic cell vaccine given intradermally at weeks 3, 6, 9, 12, 15 and 24.

SUMMARY:
Background:

- Few studies or literature are available about the long-term safety of repeated peptide vaccinations in people over a period of time. Long-term vaccination may be needed to control tumors. Researchers gave a group of men a series of vaccine injections over 2 years. Now they want to give those same men the new version of the vaccine. They want to see if it produces different types of immune responses and also ensure that repeated vaccinations are safe.

Objectives:

- To find out the long-term safety of repeated T-cell receptor alternate reading frame protein (TARP) peptide vaccinations.

Eligibility:

- Men who took part in National Cancer Institute (NCI) protocol 09-C-0139.

Design:

* Participants will be screened with blood tests, scans, physical exam, medical history, and an evaluation of how well they perform everyday activities.
* Participants will have apheresis. Blood will be removed with a needle from one arm. A machine will separate the white blood cells. The blood, minus the white cells, will be returned through a needle in the other arm.
* Participants will have 14 visits. At each visit, they will have a physical exam and blood tests. They will discuss any side effects.
* Participants will get vaccine injections at weeks 3, 6, 9, 12, 15, and 24. The vaccine will be made from the participants own cells.
* Participants will get a Vaccine Report Card to complete after receiving vaccine.
* The study lasts 96 weeks.

DETAILED DESCRIPTION:
TARP

* T-cell receptor gamma alternate reading frame protein (TARP) is an amino acid protein expressed by both normal and malignant prostate cancer tissue; 95% of prostate cancer specimens are positive for TARP expression. TARP is highly expressed in prostate cancers of all Gleason types, in primary as well as metastatic disease, and in hormone sensitive and castrate resistant prostate cancer. Therefore, TARP is an ideal tumor antigen target for a vaccine.
* A prospective, randomized pilot study of 1st generation TARP Peptide vaccination National Cancer Institute (NCI 09-C- 0139) utilizing TARP WT 27-35 and EE29-37-9V peptides was conducted in HLAA* 0201positive men with stage D0 prostate cancer prostate specific-antigen (PSA) biochemical recurrence) and a PSA doubling time (PSADT) of greater than or equal to 3 months and less than or equal to 15 months. TARP vaccination was found to be immunogenic, safe and well tolerated, with adverse events limited to injection site reactions less than or equal to Grade 2. TARP vaccination was also associated with a decreased slope log PSA compared to pre-vaccination baseline in 72% of subjects reaching 24 weeks and 74% reaching 48 weeks (p=0.0012 and p=0.0004 for overall changes in slope log PSA, respectively); TARP vaccination also resulted in a 50% decrease in calculated tumor growth rate constant: prevaccine g = 0.0042/day, post-vaccine g = 0.0021/day (p=0.003); TARP-specific IFN- >= enzyme-linked immunosorbent spot (ELISPOT) responses were detected in the majority of subjects but did not correlate with decreases in slope log (PSA).

Multi-Epitope (ME) TARP Vaccine

* The vaccine platform includes the original two 9-mer HLA-A*0201 binding TARP peptide epitopes (WT27-35 and EE29-37-9V) utilized in NCI 09-C-0139 as well as an additional five 20-mer TARP peptides overlapping by 10 amino acids for a total of 7 peptides that span the amino acid sequence of the entire TARP protein.
* The advantage of this multi-epitope TARP peptide vaccine platform is that the overlapping epitopes cover the entire TARP protein, resulting in potential for induction of a multi-valent anti-TARP response. In addition, these longer synthetic peptides include TARP-specific MHC class II CD4 T lymphocytes (CD4+ T) cell helper epitopes that will allow generation of better cyctotoxic T cells (CD8+ T) cell responses with improved functional avidity and longevity as well as humoral anti-TARP antibody responses.

Study Objectives

Primary Objective:

-To assess the long-term safety of repeated TARP peptide vaccination following the use of a 1st generation bivalent (09-C-0139) and a 2nd generation ME TARP peptide vaccine. Specifically, to document if less than 10% of enrolled patients experience a vaccine-related Grade 3 adverse event (local injection site reactions or systemic reactions).

Eligibility Criteria All Patients

* Males greater than or equal to 18 years of age with histologically confirmed adenocarcinoma of the prostate.
* Prior enrollment in NCI protocol 09-C-0139 with receipt of at least 5 doses of TARP peptide vaccine (i.e. completion of primary vaccination series).
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-1 and life expectancy greater than or equal to 1 year.
* Hemoglobin greater than or equal to 10.0 gm/dL, white blood cell (WBC) greater than or equal to 2,500/mm^3, ALC greater than or equal to 500/ mm^3, absolute neutrophil count (ANC) greater than or equal to 1,000/mm^3, platelet

count greater than or equal to 100,000/mm^3, and prothrombin time (PT)/partial thromboplastin time (PTT) less than or equal to 1.5X upper limit of normal (ULN) unless receiving clinically indicated anticoagulant therapy; serum glutamate-pyruvate transaminase (SGPT)/serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5X ULN, total bilirubin less than or equal to 1.5X ULN; creatinine less than or equal to 1.5X ULN and estimated glomerular filtration rate (eGFR) greater than or equal to 60 ml/min.

* Hepatitis B and C negative (unless the result is consistent with prior vaccination or prior infection with full recovery); human immunodeficiency virus (HIV) negative.
* No use of investigational agents within 4 weeks of study enrollment or use of immunosuppressive or immunomodulating agents within 8 weeks of study entry.
* Standard of care medical management of current prostate cancer disease status by the patients local oncologist e.g., androgen deprivation therapy is allowed.
* Must be able/willing to adhere to protocol requirements and vaccination timeline.

Exclusion Criteria All Patients

* Patients with active infection or other significant or uncontrolled medical illness. Patients with a remote history of asthma or active mild asthma may participate.
* Patients on immunosuppressive therapy including systemic corticosteroid therapy for any reason. Patients receiving inhaled or topical corticosteroids may participate.
* Patients who, in the opinion of the Principal Investigator, have significant medical or psychosocial problems that warrant exclusion.

Study Design

* Open label, prospective, non-randomized, long-term follow-up pilot study of 96 weeks to assess the long-term safety of repeated TARP vaccination in patients that have already received the first generation TARP vaccine. Sample size: N equals 40 maximum.
* All patients will undergo an 18L apheresis for mononuclear cell collection at Week 0.
* All patients will receive a total of 6 doses of autologous ME TARP peptide dendritic cell (DC) vaccine: 20x10^6 viable cells/dose) delivered intradermally at Weeks 3, 6, 9, 12, 15, and 24.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males greater than or equal to 18 years of age with histologically confirmed adenocarcinoma of the prostate.
* Prior enrollment in National Cancer Institute (NCI) protocol 09-C-0139 with receipt of at least 5 doses of T cell receptor gamma alternate reading frame protein (TARP) peptide vaccine (i.e. completion of primary vaccination series).
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-1, life expectancy of greater than or equal to 1 year.
* Hemoglobin greater than or equal to 10.0 gm/dL, white blood cell (WBC) greater than or equal to 2,500/mm^3, absolute lymphocyte count (ALC) greater than or equal to 500/mm^3, absolute neutrophil count (ANC) greater than or equal to 1,000/mm^3, platelet count greater than or equal to 100,000/mm^3.
* Prothrombin time (PT)/partial thromboplastin time (PTT) less than or equal to 1.5X upper limit of normal (ULN) unless receiving clinically indicated anticoagulant therapy.
* Serum glutamic-oxaloacetic transaminase (SGOT)/serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5X ULN, total bilirubin less than or equal to 1.5X ULN, creatinine (Cr) less than or equal to 1.5X ULN, estimated glomerular filtration rate (eGFR) greater than or equal to 60 ml/min.
* Hepatitis B and C negative, unless the result is consistent with prior vaccination or prior infection with full recovery.
* Human immunodeficiency virus (HIV) negative
* No use of investigational agents within 4 weeks of study enrollment or use of immunosuppressive or immunomodulating agents (including Intravenous immune globulin (IVIG) within 8 weeks of study entry. Note: Use of topical, inhaled and intranasal steroid therapy is permitted.
* Greater than or equal to 6 weeks since the receipt of chemotherapy or radiation therapy.
* Standard of care medical management of current prostate cancer disease status by the patients local oncologist, e.g., androgen deprivation therapy is allowed.
* Able to understand and provide Informed Consent.
* Must be able and willing to adhere to protocol requirements, visits and vaccination timeline.

EXCLUSION CRITERIA:

* Patients with a second malignancy requiring active treatment.
* Patients with an active infection.
* Patients on immunosuppressive therapy including:

  --Systemic corticosteroid therapy for any reason. Patients receiving inhaled, intranasal or topical corticosteroids may participate.
* Other significant or uncontrolled medical illness. Patients with a remote history of or active mild asthma may participate.
* Patients who, in the opinion of the Principal Investigator, have significant medical or psychosocial problems that warrant exclusion including:

  * Other serious non-malignancy-associated medical conditions that may be expected to limit life expectancy to less than 2 years.
  * Any condition- medical, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung M Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0076.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Started | 14
Completed | 8
Not Completed | 6
Not completed — Switched to alternative therapy | 1
Not completed — Refused further treatment | 1
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.14 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3 Adverse Events (AEs) Probably Related to the Vaccine Treatment
Description: The number of Grade 3 adverse events probably related to the vaccine treatment. Adverse events were measured using the Common Terminology Criteria for Adverse Events (CTCAE v.4.0). Grade 3 is severe.
Time Frame: Up to 30 days after week 24 vaccination
Measure: Number; unit: Adverse events
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Number analyzed (Participants) | 14
Adverse events | 1

2. Secondary Outcome: Change in Slope Log PSA From Pre-study Baseline (-12 Months to Entry on the Current Study) to the Change in Slope Log PSA at Weeks 3-24 and 3-48 Post Multi-Epitope (ME) T-cell Receptor Alternate Reading Frame Protein (TARP) Vaccination
Description: "PSA slope log" was calculated using Memorial Sloan Kettering Cancer Center Prostate Cancer Nomograms (http://nomograms.mskcc.org/Prostate/PsaDoublingTime.aspx) Slope log represents the speed of change of a series of values. Thus, it is reported without any units as it is with a concept of ratio. The clinical meaning of PSA slope change would be decrease or increase of the "speed (velocity)" of changes in PSA, not the changes in PSA values. Decreasing PSA slope after the investigational treatment would mean the PSA rise is slower than pre-treatment baseline. Lowered PSA slope has been reported to show a relationship with was reported as related to improved outcomes.
Time Frame: Weeks 3-24 minus baseline, and Weeks 3-48 minus baseline
Population: Study participants who were in biochemically recurrent prostate cancer and not exposed to androgen deprivation therapy for the management of prostate cancer were evaluable for this endpoint.
Measure: Median (Full Range); unit: Slope log
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Number analyzed (Participants) | 6
Slope log
  Weeks 3-24 | -0.00 [-0.09 to 0.10]
  Weeks 3-48: number analyzed (Participants) | 5
  Weeks 3-48 | -0.01 [-0.04 to 0.08]

3. Secondary Outcome: Change in Slope Log Prostate Specific-antigen (PSA) Versus the Same Change in Slope Log PSA Parameters Following 1st Generation T-cell Receptor Alternate Reading Frame Protein (TARP) Vaccination on Protocol 09-C-0139
Description: Participants slope log on study 09C0139 are compared with the slope log values for the same participants after receiving the updated ME-TARP vaccines on the current protocol 15C0076 in participants who were not treated with androgen deprivation. PSA slope log was calculated using Memorial Sloan Kettering Cancer Center Prostate Cancer Nomograms (http://nomograms.mskcc.org/Prostate/PsaDoublingTime.aspx) Slope log represents the speed of change of a series of values. Thus, it is reported without any units as it is with a concept of ratio. The clinical meaning of PSA slope change would be decrease or increase of the "speed (velocity)" of changes in PSA, not the changes in PSA values. Decreasing PSA slope after the investigational treatment would mean the PSA rise is slower than pre-treatment baseline. Lowered PSA slope has been reported to show a relationship with was reported as related to improved outcomes.
Time Frame: Weeks 3-24 minus baseline, and Weeks 3-48 minus baseline
Population: The participants who were evaluable for Memorial Sloan Kettering Cancer Center Prostate Cancer Nomograms are reported for this outcome measure.
Measure: Median (Full Range); unit: Slope log
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Number analyzed (Participants) | 6
Slope log
  PSA slope log of the participants while on previous study 09C0139 at Weeks 3-24 | -0.06 [-0.175 to 0.018]
  PSA slope log of the participants while on current study 15C0076 at Weeks 3-24 | -0.00 [-0.09 to 0.10]
  PSA slope log of the participants while on previous study 09C0139 at Weeks 3-48: number analyzed (Participants) | 5
  PSA slope log of the participants while on previous study 09C0139 at Weeks 3-48 | -0.03 [-0.116 to 0.012]
  PSA slope log of the participants while on current study 15C0076 at Weeks 3-48: number analyzed (Participants) | 5
  PSA slope log of the participants while on current study 15C0076 at Weeks 3-48 | -0.01 [-0.04 to 0.08]

4. Secondary Outcome: Number of Participants With Reactivity to WT27-35 and EE29-37-9V T-cell Receptor Alternate Reading Frame Protein (TARP) Peptides
Description: Measure of activity to WT27-35 and EE29-37-9V TARP peptides was done by interferon (IFN)-gamma enzyme-linked immunosorbent spot (ELISPOT) assay. Positivity was defined by higher counts of spot counts than the counts in negative controls. and reactivity defined by higher spot counts than the negative controls.
Time Frame: Week 24 and Week 48 following immunization with the 2nd generation Multi-Epitope (ME) TARP
Population: 13/14 participants were evaluable for this outcome measure. Week 48 was not done due to issues in laboratory resources: samples were available in very limited number of participants and assay was not done (data not collected). As the samples were too low, the cost/resources needed to analyze week 48 were prohibitive funding wise considering the limited information to be generated with a small sample size.
Measure: Count of Participants; unit: Participants
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Number analyzed (Participants) | 13
Participants
  Week 24 Reactive to TARP WT27-35 | 5
  Week 24 Reactive to TARP EE29-37 | 9
  Week 24 Reactive to Both Peptides | 5
  Week 24 Not Reactive to Any of the Peptides | 4
  Week 48: number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Positive for T-cell Receptor Alternate Reading Frame Protein (TARP) WT27-35 and EE29-37-9V Peptide Reactivity to That of the 1st Generation TARP Vaccine in the Same Individuals on Protocol 09-C-0139 (NCT00972309) and 15-C0076
Description: Number of participants positive for WT27-35 and EE29-37-9V TARP peptide interferon (IFN)-gamma enzyme-linked immunosorbent spot (ELISPOT) reactivity. Positivity was defined by higher counts of spot counts than the counts in negative controls.
Time Frame: Week 24 and 48 following Multi-Epitope (ME) TARP vaccination
Population: 13/14 participants were evaluable for this outcome measure. Week 48 not done due to issues in laboratory resources: Week 48 was not done due to issues in laboratory resources: samples were available in very limited number of participants and assay was not done (data not collected). As the samples were too low, the cost/resources needed to analyze week 48 were prohibitive funding wise considering the limited information to be generated with a small sample size.
Measure: Count of Participants; unit: Participants
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Number analyzed (Participants) | 13
Participants
  Week 24 Positive for WT27-35 Peptide in 09C0139 | 7
  Week 24 Positive for WT27-35 Peptide in 15C0076 | 6
  Week 24 Positive for TARP EE29-37 Peptide in 09C0139 | 8
  Week 24 Positive for TARP EE29-37 Peptide in 015C0076 | 8
  Week 48: number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 82 months and 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
Number analyzed (Participants) | 14
Participants | 13

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 82 months and 6 days.
Arm/Group | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations (N=14)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term T-cell Receptor Alternate Reading Frame Protein (TARP) Peptide Vaccinations (N=14)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood and lymphatic system disorders - Other, red streak in right arm (Blood and lymphatic system disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (5)
Fever (General disorders) | 1 (2)
Flu like symptoms (General disorders) | 1 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, tooth chip (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (7)
Injection site reaction (General disorders) | 13 (127)
Insomnia (Psychiatric disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — squamous cell; Left shin
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (3)
Skin and subcutaneous tissue disorders - Other, Soft nodule on the right temporal region, non tender (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, chronically dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, genital herpes lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, lump under right 1st toe nail (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT02362464/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Addendeum Consent (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02362464/ICF_001.pdf
  • Informed Consent Form: Cohort Affected Participant Consent (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02362464/ICF_002.pdf